CLINICAL TRIAL: NCT03751891
Title: Quality Control of CE-Certified Phonak Hearing Aids - Sonova2018_05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2018_05
Record Dates: First submitted 2018-09-14; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant masking was only done for laboratory measurements. For home trial testing no masking was done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phonak Audéo B90-Direct (Experimental): The Phonak Audéo B90-Direct is the most recent Receiver-in-the-canal Hearing aid with direct connectivity functionality from Phonak which will be fitted to the participants individual Hearing loss.
  Interventions: Device: Phonak Audéo B90-Direct
- HearingAid_A (Active Comparator): HearingAid_A is the most recent Receiver-in-the-canal Hearing aid with direct connectivity functionality from manufacturer_A which will be fitted to the participants individual Hearing loss.
  Interventions: Device: HearingAid_A
- HearingAid_B (Active Comparator): HearingAid_B is the most recent Receiver-in-the-canal Hearing aid with direct connectivity functionality from manufacturer_B which will be fitted to the participants individual Hearing loss.
  Interventions: Device: HearingAid_B

INTERVENTIONS:
Device: Phonak Audéo B90-Direct — The Phonak Audéo B90-Direct is the most recent Receiver-in-the-canal Hearing aid from Phonak which will be fitted to the participants individual Hearing loss.
  Arms: Phonak Audéo B90-Direct
Device: HearingAid_A — HearingAid_A is the most recent Receiver-in-the-canal Hearing aid from manufacturer_A which will be fitted to the participants individual Hearing loss.
  Arms: HearingAid_A
Device: HearingAid_B — HearingAid_B is the most recent Receiver-in-the-canal Hearing aid from manufacturer_B which will be fitted to the participants individual Hearing loss.
  Arms: HearingAid_B

SUMMARY:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Phonak Hearing Systems undergo a final quality control in terms of clinical trials. This is a validation study, investigating optimized algorithms, features, functions and wearing comfort. This will be a clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

DETAILED DESCRIPTION:
In this study a comparison with a CE-labeled Phonak Receiver-in-the-canal (RIC) device (active comparator) and two CE-labeled competitor devices (RIC) is done. All study devices contain direct connectivity functionality which will be compared in terms of streamed Audio quality, streaming stability and Usability preferences of all available functions and features. This will be a clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years, mild to moderate Hearing loss) without hearing aid experience
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* willingness to wear Receiver in the canal hearing aids
* Informed Consent as documented by signature
* owning an iPhone 6 or higher

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Known psychological problems
* Central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the speech intelligibiltity of phone calls via direct streaming | 6 weeks
  The primary outcome meaurement of this study is the comparison of Phonak's direct connectivity solution against two competitors in terms of subjective speech intelligibility of streamed audio signals via smartphone. The subjective speech intelligibilty will be measured via interview (sound quality rating, satisfaction rating of speech intelligibility) from far-end talker and near-end talker.

SECONDARY OUTCOMES:
Investigation of Bluetooth Connection losses between Hearing Aid and smart phone during a phone call (number of reported interruptions during a phone call which will be streamed via bluetooth from Smartphone to Hearing Aid) | 6 weeks
  The secondary outcome measurement of this study is to investigate the number of (Bluetooth-) Connection losses between Hearing Aid and Smartphone during a phone call stream. The bluetooth connection losses will be investigated by counting the reported interruptions of a streamed phone call between smartphone and Hearing Aid in relation to the amount of conducted phone calls during two weeks of home trial for the investigational device and the comparative devices.

OTHER OUTCOMES:
Comparison of the subjective Sound Quality rating of TV-Audiostream via direct connectivity | 6 weeks
  Another outcome measurement of this study is the comparison of streamed audio signals from TV in terms of sound quality (measured via satisfaction rating).
Comparison of the Usability of remote controls via direct connectivity | 6 weeks
  Another outcome measurement of this study is the comparison of the usability of a remote control via interview during and after home trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland